CLINICAL TRIAL: NCT04116073
Title: A Phase II Trial of INCMGA00012 in Patients With Previously Treated Unresectable or Metastatic Adenosquamous Pancreatic or Ampullary Cancer
Brief Title: INCMGA00012 in Patients With Previously Treated Unresectable or Metastatic Adenosquamous Pancreatic or Ampullary Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Incyte Corporation (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J19106; IRB00224849 (Other: Johns Hopkins Medical Institution); P50CA062924 (NIH)
Record Dates: First submitted 2019-10-03; First posted 2019-10-04 (Actual); Results first posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Pancreatic Cancer Non-resectable; Pancreatic Cancer Metastatic
Keywords: Antibody; Anti-PD-1; Human monoclonal immunoglobulin antibody; Immunotherapy; INCMGA00012 (anti-PD-1 antibody); Anti-PD-1 antibody (MGA012); Metastatic adenosquamous pancreatic cancer; Unresectable adenosquamous pancreatic cancer; Adenosquamous pancreatic cancer; Programmed cell death protein 1 (PD-1); Programmed death-ligand 1 (PD-L1)
MeSH Terms: conditions — Parkinson Disease 4, Autosomal Dominant Lewy Body

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- INCMGA00012 (PD-1 antibody) (Experimental): All participants received the interventional study drug; INCMGA00012.
  Interventions: Drug: INCMGA00012 (PD-1 antibody)

INTERVENTIONS:
Drug: INCMGA00012 (PD-1 antibody) — INCMGA00012 (PD-1 antibody): 500 mg, 30 min IV infusion on Day 1 of each cycle (every 28 days)
  Other Names: MGA012

SUMMARY:
Phase 2 study to evaluate the clinical activity of INCMGA00012 in patients with Unresectable or metastatic Adenosquamous Pancreatic or Ampullary Cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Have histologically or cytologically - proven adenosquamous carcinoma of the pancreas or ampulla.
* Has unresectable or metastatic measurable disease.
* Has received (or been intolerant to or ineligible for) at least 1 prior line of cytotoxic chemotherapy and received no more than 2 prior systemic treatments.
* Presence of at least one lesion with measurable disease.
* Accept to have a tumor biopsy of an accessible lesion at baseline and on treatment.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* If HIV-positive, then all of the following criteria must also be met: cluster of differentiation (CD) 4+ count ≥ 350/μL, undetectable viral load, and receiving highly active antiretroviral therapy.
* Life expectancy of greater than 3 months.
* Patients must have adequate organ and marrow function defined by study-specified laboratory tests prior to initial study drug.
* Woman of childbearing potential must have a negative pregnancy test and follow contraceptive guidelines as defined per protocol.
* Men must use acceptable form of birth control while on study.
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria

* Known history or evidence of brain metastases.
* Has had chemotherapy, radiation, or biological cancer therapy within 14 days prior to the first dose of study drug.
* Has received an investigational agent or used an investigational device within 28 days of the first dose of study drug.
* Expected to require any other form of systemic or localized antineoplastic therapy while on study.
* Has had major surgery within 28 days of dosing of investigational agent, excluding minor procedures.
* Has received a live vaccine within 28 days prior to the first dose of study drug.
* Prior treatment with immunotherapy agents (including, anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA4, anti-OX40 and LAG-3 antibodies)
* Have used any systemic steroids within 14 days of study treatment.
* Hypersensitivity reaction to any monoclonal antibody.
* Evidence of clinical or radiographic ascites.
* Have clinically significant and/or malignant pleural effusion.
* Uncontrolled intercurrent illness including, but not limited to, uncontrolled infection, symptomatic congestive heart failure, unstable angina, cardiac arrhythmia, metastatic cancer, or psychiatric illness/social situations that would limit compliance with study requirements.
* History of autoimmune disease requiring systemic immunosuppression within the last 2 years.
* Presence of any tissue or organ allograft, regardless of need for immunosuppression, including corneal allograft. Patients with a history of allogeneic hematopoeitic stem cell transplant will be excluded.
* All toxicities attributed to prior anti-cancer therapy other than alopecia and fatigue must have resolved to a grade 1 or baseline before administration of study drug.
* Infection with Hepatitis A, B or C.
* Patient has a pulse oximetry of <92% on room air.
* Patient is on supplemental home oxygen.
* Has an unhealed surgical wound or ulcer, or a bone fracture considered non-healing.
* Patient has clinically significant heart disease.
* Patient is, at the time of signing informed consent, a regular user (including "recreational use") of any illicit drugs or other substance abuse.
* Unwilling or unable to follow the study schedule for any reason.
* Patient has history of non-infectious pneumonitis.
* Serum albumin level less than 2.8 g/dL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-04-09 (Actual); Primary Completion 2024-08-06 (Actual); Study Completion 2024-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nilofer Azad, MD, Principal Investigator — Johns Hopkins Medical Institution
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | INCMGA00012 (PD-1 Antibody)
Started (Started=enrolled on study.) | 25
Completed (Completed= received at least one dose of the study drug.) | 22
Not Completed | 3
Not completed — Withdrawal by Subject | 2
Not completed — failed to maintained eligibility | 1

BASELINE CHARACTERISTICS:
Population: Participants with data collected.
Arm/Group | INCMGA00012 (PD-1 Antibody)
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 18
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — The ECOG scale measures performance status, with scores ranging from 0-5; 0= fully active, performs without restriction, 1= can ambulate, but restricted in physically strenuous activity, 2= ambulatory and capable of self-care, but unable to work, active for >50% of waking hours, 3= limited self-care, confined to bed or chair for >50% of waking hours, 4= completely disabled, totally confined to bed/chair, 5= deceased.
  Participants
    ECOG 0 | 6
    ECOG 1 | 16

OUTCOME MEASURES:

1. Primary Outcome: Disease Control Rate (DCR) at 4 Months Using RECIST 1.1
Description: Disease control rate (DCR) is defined as the proportion of subjects with complete response, partial response and stable disease based on RECIST 1.1 criteria. CR = disappearance of all target lesions, PR is =>30% decrease in sum of diameters of target lesions. SD=Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. Subjects who discontinue due to toxicity prior to post-baseline tumor assessments will be evaluable and considered treatment failures.
Time Frame: 4 months
Population: One subject didnt have a follow up scan after receiving a dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | INCMGA00012 (PD-1 Antibody)
Number analyzed (Participants) | 21
Participants | 2

2. Secondary Outcome: Objective Response Rate (ORR) Using RECIST 1.1.
Description: ORR is defined as the proportion subjects with partial response (PR) or complete response (CR) according to RECIST 1.1. Subjects who discontinue due to toxicity or clinical progression prior to post-baseline tumor assessments will be considered as non-responders
Time Frame: 4 years
Population: One subject didnt have a follow up scan after receiving a dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | INCMGA00012 (PD-1 Antibody)
Number analyzed (Participants) | 21
Participants | 0

3. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) is defined as the number of months from the first dose of retifanlimab to radiographic disease progression (PD or relapse from CR as assessed using RECIST 1.1 criteria), documented clinical progression as assessed by the treating provider, or death due to any cause. PFS will be censored at the date of the last scan for subjects without documentation of disease progression at the time of analysis.
Time Frame: 34 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | INCMGA00012 (PD-1 Antibody)
Number analyzed (Participants) | 22
months | 1.8 [1.6 to 2]

4. Secondary Outcome: Grade 3 and Higher Study Drug-related Toxicities.
Description: Number of participants experiencing study drug-related adverse events Grade 3 or higher as defined by CTCAE v5.0.
Time Frame: 26 months
Measure: Count of Participants; unit: Participants
Arm/Group | INCMGA00012 (PD-1 Antibody)
Number analyzed (Participants) | 22
Participants
  Any grade 3 and higher related AE | 3
  ALT increased | 2
  AST increased | 1
  Hypophosphatemia | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected for up to 26 months. Subjects were followed for survival for up 56 months.
Arm/Group | INCMGA00012 (PD-1 Antibody)
All-Cause Mortality (participants affected / at risk) | 17/25
Serious Adverse Events (participants affected / at risk) | 9/25
Other Adverse Events (participants affected / at risk) | 21/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | INCMGA00012 (PD-1 Antibody) (N=25)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 1 (1)
Aspartate Aminotransferase Increased (Investigations) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Bile Duct Stenosis (Hepatobiliary disorders) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 1 (1)
Disease Progression (General disorders) | 5 (5)
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Lung Infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | INCMGA00012 (PD-1 Antibody) (N=25)
Anemia (Blood and lymphatic system disorders) | 4 (10)
Hypothyroidism (Endocrine disorders) | 3 (3)
Abdominal Pain (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Chills (General disorders) | 2 (2)
Edema Limbs (General disorders) | 4 (4)
Fatigue (General disorders) | 8 (8)
Fever (General disorders) | 3 (3)
Thrush (Infections and infestations) | 4 (4)
Urinary Tract Infection (Infections and infestations) | 2 (4)
Bruising (Injury, poisoning and procedural complications) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 3 (3)
Alanine Aminotransferase Increased (Investigations) | 2 (6)
Alkaline Phosphatase Increased (Investigations) | 3 (4)
Aspartate Aminotransferase Increased (Injury, poisoning and procedural complications) | 3 (5)
Lymphocyte Count Decreased (Injury, poisoning and procedural complications) | 2 (3)
Weight Gain (Investigations) | 3 (3)
Weight Loss (Investigations) | 8 (11)
Anorexia (Metabolism and nutrition disorders) | 3 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (4)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Headache (Nervous system disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (4)
Rash Acneiform (Skin and subcutaneous tissue disorders) | 2 (2)
Thromboembolic Event (Vascular disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-20): https://cdn.clinicaltrials.gov/large-docs/73/NCT04116073/Prot_SAP_000.pdf